CLINICAL TRIAL: NCT01012427
Title: Percutaneous Renal Tumor Cryoablation Followed by Biopsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-108
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Renal Cancer
Keywords: Kidney; Cryoablation; 09-108
MeSH Terms: conditions — Kidney Neoplasms

ARMS (1):
- Patients with 3.0 cm or smaller renal cancer (Experimental): The interventions in this study are part of clinical care and include percutaneous image-guided biopsy, percutaneous renal tumor cryoablation, CT/MR imaging of the ablation bed, and repeat pathologic sampling of the tumor bed with percutaneous biopsy. The cryoablation is done as the therapeutic intervention in patients with small renal cancer. The CT/MR imaging is done to evaluate the treatment for residual disease after the ablation. The repeat biopsy (e.g. three cores) is done to confirm that the neoplasm has been eradicated. These patients have continued imaging, and if necessary, percutaneous biopsy to ensure no recurrent disease.
  Interventions: Procedure: percutaneous cryoablation

INTERVENTIONS:
Procedure: percutaneous cryoablation — All patients will have percutaneous image guided core biopsies of the treatment site and CT or MR imaging at approximately 5-7 months following the cryoablation. They will have repeat imaging every 5-7 months for a period of two years, and if there is evidence of recurrence (ablation zone increase > 5 mm or increased enhancement 15 HU), then repeat biopsy will be obtained. Imaging follow-up past the two year point will be at the discretion of the patient's physicians.

SUMMARY:
This study is being done to test how effective cryoablation is in killing cancer cells. Cryoablation uses freezing temperatures to treat cancer. Cryoablation works by creating freezing temperatures within a needle probe. When this probe is inserted into a cancer, the freezing temperatures are used to try and kill the cancer. Unfortunately, the investigators don't know how well cryoablation works at destroying the cancer. This study will allow us to check to see how well cryoablation works for kidney cancers. After the investigators destroy the kidney cancers using cryoablation, the investigators will followup with you every 5-7 months to make sure the cryoablation worked and that the cancer was destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one renal cancer smaller than or equal to 3.0 cm
* Adequate baseline imaging studies (CT/MRI) within 8 weeks of treatment or as clinically indicated.
* The following laboratory results should be within the following limits within the last 30 days prior to study day 1. Repeat blood work will be necessary if too much time has elapsed prior to the interventions.:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Serum bilirubin ≤ 2.0 mg/dL
* Aspartate aminotransaminase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Serum creatinine ≤ 2.0 mg/dL
* GFR >30 mL/min/m2
* International Normalized Ratio < 1.5 (INR)
* Partial Thromboplastin Time (PTT) <45 seconds
* Recovered from toxicity of any prior therapy
* Tumor accessible to probe placement without risk to adjacent critical structures.
* Tumor visible on non-contrast CT
* Patient willing and able to undergo imaging and percutaneous biopsy at 5-7 month intervals for 2 years and then at the discretion of the patient's physicians.

Exclusion Criteria:

* Intercurrent medical condition that renders the patient ineligible for cryoablation
* Women who are pregnant or breastfeeding.
* Tumor less than 5 mm to the renal pelvis, main renal vessel, ureter, or other vital structure
* Contraindication to MRI in patients in which it is required.
* Coagulopathy as defined above (Inclusion Criteria).
* Patients unwilling to return for follow-up biopsy and imaging.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy rate after percutaneous renal cryoablation. | 2 years

SECONDARY OUTCOMES:
To determine the complication rate of percutaneous renal tumor cryoablation. | 2 years
To correlate post-treatment imaging parameters of CT/MR with therapeutic cryoablation success. | 2 years
To assess the glomerular filtration rate changes associated with percutaneous renal cryoablation. | 2 years
To investigate predictors of efficacy after cryoablation. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Solomon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm